CLINICAL TRIAL: NCT03642028
Title: Suvorexant: A Dual Orexin Receptor Antagonist for Treating Sleep Disturbance inPosttraumatic Stress
Brief Title: Suvorexant: A Dual Orexin Receptor Antagonist for Treating Sleep Disturbance in Posttraumatic Stress
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-009-17F; 1I01CX001814-01 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Sleep Initiation and Maintenance Disorders; Stress Disorders, Posttraumatic
Keywords: Sleep Initiation and Maintenance Disorders; Stress Disorders, Posttraumatic; Suvorexant; Veterans
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: The investigators propose a multi-site parallel group, randomized, double-blind, placebo-controlled Phase IV clinical trial to test the efficacy and safety of suvorexant on trauma-related sleep disturbance and PTSD symptoms in Veterans. The investigators will use a flexible dose design of suvorexant with a 2-week titration followed by a 10-week steady-dose phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blind will be maintained through completion of the entire study at all sites and will only be broken once data are cleaned to an acceptable level of quality, except for medical necessity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant (Experimental): Suvorexant is a dual orexin receptor antagonist that is FDA approved to treat insomnia.
  Interventions: Drug: Suvorexant
- Identical Placebo (Placebo Comparator): Visibly matched, equally weighted placebo tablets. In addition to matching in appearance and weight, they will have identical packaging and labeling as randomized, blinded study medication.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Suvorexant — Suvorexant, a dual orexin receptor antagonist, is the first in a new class of drugs with great promise of addressing insomnia in Veterans with PTSD. Suvorexant targets the orexin neuropeptide system and has been shown to be highly successful in treating insomnia.
  Other Names: Belsomra
  Arms: Suvorexant
Other: Placebo — Visibly matched, equally weighted placebo tablets. In addition to matching in appearance and weight, they will have identical packaging and labeling as randomized, blinded study medication.
  Arms: Identical Placebo

SUMMARY:
Post-traumatic stress disorder (PTSD) is a common consequence of combat that can result in trauma-related hyperarousal and sleep disturbances. Poor sleep, one of the most common complaints in Veterans with PTSD, can be distressing, impair concentration and memory, and contribute to physical health conditions, such as metabolic syndrome, inflammation, and cardiovascular disease. The orexin neuropeptide system underlies both sleep and stress reactivity. Suvorexant, a drug that reduces orexin, improves sleep in civilians, but has not yet been tested in Veterans with PTSD. This study will test whether suvorexant can improve sleep disturbances and PTSD symptoms in Veterans. Suvorexant may benefit Veterans by improving sleep quickly while also reducing PTSD symptoms over the long term, and with fewer side effects that were common in previous medications used to treat these conditions. Improving Veterans' sleep and PTSD symptoms could lead to better emotional and physical well-being, quality of life, relationships, and functioning.

DETAILED DESCRIPTION:
The investigators propose a multi-site parallel group, randomized, double-blind, placebo-controlled Phase IV clinical trial to test the efficacy and safety of suvorexant on trauma-related sleep disturbance and PTSD symptoms in Veterans. The investigators will use a flexible dose design of suvorexant with a 2-week titration followed by a 10-week steady-dose phase. The investigators predict that suvorexant, as compared to placebo, will result in a greater decrease in insomnia on the Insomnia Severity Index (ISI) over the 12-week trial. The investigators also predict that suvorexant, as compared to placebo, will result in a greater reduction in non-sleep PTSD symptoms in the Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSMV) (CAPS-5) over the 12-week trial. Secondarily, the investigators will examine potential objectively measured wrist actigraphy as a biological mechanism of clinical improvement with as well as concomitant effects on PTSD-related nightmares using the Pittsburgh Sleep Quality Index-PTSD addendum (PSQI-A). Pending a significant effect of suvorexant on PTSD, the investigators will perform exploratory analyses to evaluate whether sleep improvement mediates the effect of suvorexant on PTSD symptoms. The investigators will also examine safety and tolerability of suvorexant compared to placebo (including depression, mood, vigor, suicidality, and daytime somnolence, psychomotor vigilance, and functional disability). Results from this study will provide substantive rationale for the use of Suvorexant in the treatment of Veterans with these concerns. This study will be the first to examine a selective orexin-receptor antagonist in a Veteran sample with PTSD. Suvorexant is an accessible, non-stigmatized medication whose use and safety has been well-established in non-mental-health settings. It has outstanding promise for treating common and distressing symptoms in Veterans as well as civilians with trauma-related sleep disturbance and PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women, age range of 18 to 75, with a history of US military service, capable of reading and understanding English, and able to provide written informed consent
* Criterion A event meets DSM-5 criteria
* PTSD symptoms >3 months duration as indexed by a CAPS-5 12 and a partial PTSD diagnosis at screening
* Insomnia indicated by an ISI score > 14
* Subjects on non-exclusionary medications must be on a stable dose for at least 4 weeks prior to randomization, which includes the Selective Serotonin Reuptake Inhibitors (SSRIs) e.g.:

  * Sertraline
  * Paroxetine
  * Fluoxetine
  * Fluvoxamine
  * Citalopram
  * Escitalopram
* Serotonin-norepinephrine reuptake inhibitors (SNRIs), e.g.:

  * Desvenlafaxine
  * Duloxetine
  * Levomilnacipran
  * Venlafaxine
* For subjects who are in psychotherapy, treatment must be stable for 6 weeks
* Women of child-bearing potential must not be pregnant or have plans for pregnancy or breastfeeding during the study and must use a medically acceptable method of birth control, e.g.:

  * oral
  * implantable
  * injectable
  * transdermal contraceptive
  * intrauterine device
  * double-barrier method
* Sleep apnea score <30; if screening indicates mild or moderate sleep apnea (score between 5 and 30), referral will be provided

Exclusion Criteria:

* DSM-5 alcohol, marijuana, and/or other drug use disorder in the last 3 months

  * Mild alcohol use not meeting criteria for moderate or severe use disorder may be allowed on a case-by-case basis
  * Mild or moderate marijuana use disorder may be allowed on a on a case-by-case basis
* Manic or psychotic episode in the last 5 years
* Exposure to trauma in the last 3 months
* Prominent suicidal or homicidal ideation or any suicidal behavior in the past 3 months on the Columbia Suicide Severity Rating Scale (C-SSRS) or increased risk of suicide that necessitates additional therapy or inpatient treatment
* Pre-existing severe sleep apnea (score >30) in the absence of adherence to effective treatment (such as CPAP or oral device) or positive screen for severe sleep apnea by type III device (score > 30)
* Neurologic disorder or systemic illness affecting CNS function
* Chronic or unstable medical illness including:

  * unstable angina
  * myocardial infarction within the past 6 months
  * congestive heart failure
  * preexisting hypotension or orthostatic hypotension
  * heart block or arrhythmia
  * chronic renal or hepatic failure
  * pancreatitis
  * severe chronic obstructive pulmonary disease
* History of severe traumatic brain injury
* Mild cognitive impairment assessed by the Montreal Cognitive Assessment
* Pregnancy, breastfeeding and/or refusal to use effective birth control (for women)
* Narcolepsy
* Previous adverse reaction to a hypnotic
* Current use of benzodiazepines, strong CYP3A inhibitors, or Digoxin

Prohibited:

* benzodiazepines
* strong CYP3A inhibitors
* Digoxin
* Furthermore, CNS depressants (e.g., benzodiazepines, opioids, alcohol) increase the risk of CNS depression when co-administered with suvorexant and will not be allowed for safety reasons.
* Since metabolism by CYP3A is the major elimination pathway for suvorexant, concomitant use of suvorexant with strong inhibitors of CYP3A (e.g., ketoconazole, itraconazole, posaconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, boceprevir, telaprevir, telithromycin and conivaptan), moderate CYP3A inhibitors (e.g., amprenavir, aprepitant, atazanavir, ciprofloxacin, diltiazem, erythromycin, fluconazole, fosamprenavir, grapefruit juice, imatinib, verapamil), or strong CYP3A inducers (e.g., rifampin, carbamazepine and phenytoin) will not be allowed.
* All concomitant medication use will be monitored and documented

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline to week 12
  The ISI is a specific index of perceived insomnia severity. Areas assessed include problems with sleep onset, sleep maintenance, and early morning awakening; dissatisfaction with sleep; interference with daily functioning; impact on quality of life; and worry about sleep problems.
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Change from baseline to week 12
  The CAPS-5 is a 30-item interview that is the gold standard assessment for PTSD. The CAPS-5 provides a dimensional and categorical measure of PTSD, and incorporates frequency and intensity of symptoms into a single severity score. The CAPS-5 will determine a threshold for PTSD severity (past week) at baseline (excluding change in item #20 falling and staying asleep). Possible scores range from 0 to 80. All trained and certified CAPS-raters will function independently and will not be involved in recruitment, study coordination, or evaluation of side effects.

SECONDARY OUTCOMES:
Wrist Actigraphy | Change from 1 week at baseline, and weeks 4, 8, and 12
  Sleep wake schedule will be monitored with wrist actigraphy (Micro Motionlogger, Ambulatory Monitoring, Inc.). The actigraph provides continuous activity data using a battery-operated wristwatch-size microprocessor that senses motion with a three axis accelerometer. High-resolution data will be down-sampled to one-minute sample intervals for conventional actigraphic sleep-wake estimation and analyzed using ActionW-2 (Ambulatory Monitoring, Inc.) software. Sleep efficiency, sleep maintenance, total sleep time and wake after sleep onset will be used as secondary measures of sleep.
Pittsburgh Sleep Quality Index-PTSD Addendum (PSQI-A) | Change in PTSD-related nightmares across the 12 week trial
  PSQI-A will be used to assess disruptive nocturnal behaviors related to PTSD, including nightmares, hot flashes and episodes of terror during sleep. Scores ranges from 0 (normal) to 21 (severe). The investigators plan to evaluate nightmares as a secondary outcome.

OTHER OUTCOMES:
Clinical Global Impression (CGI) | Change across the 12 week trial
  The Clinician and patient reports of improvement on the CGI (depression, mood, vigor, suicidality, daytime somnolence, and functional disability rating scales.) The CGI measures psychiatric treatment response by evaluating global severity of illness and change in the clinical condition over time. It consists of 3 global subscales: Severity of Illness, Global Improvement, and Efficacy Index. Item 1 is rated on a seven-point scale (1=normal to 7=extremely ill); item 2 on a seven-point scale (1=very much improved to 7=very much worse); and item 3 on a four-point scale (from 'none' to 'outweighs therapeutic effect'). The CGI will be used as a secondary measure of remission (i.e., CGI-I of 1 "very much improved" or 2 "much improved").

CONTACTS AND LOCATIONS:
Overall Officials: Sabra S Inslicht, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (4):
- United States (4):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://studypages.com/s/are-you-a-veteran-with-sleeping-problems-and-posttraumatic-stress-participate-in-a-clinical-research-study-from-home-601539/